CLINICAL TRIAL: NCT07188350
Title: Neuromuscular Electrical Stimulation of Lower Limbs in Patients Undergoing Invasive Mechanical Ventilation: Randomized Clinical Trial
Brief Title: Neuromuscular Electrical Stimulation in a Patient on Invasive Mechanical Ventilation (MOVCARE)
Acronym: MOVCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Cassiano Teixeira, Professor Doutor, Hospital Moinhos de Vento
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOVCARE2025-LB
Record Dates: First submitted 2025-07-15; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation; Critical Illness; Intensive Care Unit Patients; Muscle Weakness Condition; Neuromuscular Electrical Stimulation (NMES)
Keywords: Neuromuscular Electrical Stimulation; Physiotherapy; Mechanical Ventilation; Muscle Strength; Randomized Controlled Trial; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups in a parallel design: the control group receiving conventional physical therapy, and the intervention group receiving conventional physical therapy plus neuromuscular electrical stimulation. Both groups will be treated simultaneously during the study period.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to participant group assignment to minimize bias in outcome evaluation. Participants and care providers will be aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Physical Therapy (Active Comparator): Participants in this group will receive individualized conventional physical therapy, including progressive mobility exercises, in-bed activities (e.g., rolling, sitting at the edge of the bed), standing, transferring to a chair, walking, and respiratory therapy as clinically indicated. Treatments will be adjusted daily based on each patient's physiological status.
  Interventions: Other: Conventional Physical Therapy
- Conventional Physical Therapy + Neuromuscular Electrical Stimulation (Experimental): Participants in this group will receive the same conventional physical therapy as the control group, plus neuromuscular electrical stimulation (NMES) applied to both lower limbs once or twice daily for 20 consecutive days. NMES will be administered to the vastus lateralis, vastus medialis, tibialis anterior, hamstrings, and gastrocnemius muscles using specific parameters to produce effective muscle contractions, following a progressive stimulation protocol throughout the intervention period.
  Interventions: Other: Conventional Physical Therapy; Device: Neuromuscular Electrical Stimulation (NMES)

INTERVENTIONS:
Other: Conventional Physical Therapy — Individualized physical therapy including progressive mobility (e.g., bed exercises, sitting on the edge of the bed, standing, transfers, and ambulation) and respiratory therapy tailored to the patient's clinical condition. Delivered daily by trained professionals.
Device: Neuromuscular Electrical Stimulation (NMES) — NMES will be applied to both lower limbs once or twice daily for 20 consecutive days. Electrodes will be positioned on the vastus lateralis, vastus medialis, tibialis anterior, hamstrings, and gastrocnemius muscles. The stimulation protocol includes progressive parameters to induce visible and effective muscle contractions.
  Arms: Conventional Physical Therapy + Neuromuscular Electrical Stimulation

SUMMARY:
This clinical study aims to compare the effects of conventional physical therapy alone versus conventional physical therapy combined with neuromuscular electrical stimulation (NMES) in patients admitted to the ICU and undergoing invasive mechanical ventilation. Participants will be randomly assigned to receive either conventional physical therapy or the same therapy plus NMES applied to the lower limbs. The protocol includes muscle-specific stimulation parameters and safety criteria to postpone sessions in cases of clinical instability. The primary goal is to assess whether NMES improves muscle function and recovery in critically ill patients.

DETAILED DESCRIPTION:
This randomized clinical trial will investigate the effects of neuromuscular electrical stimulation (NMES) in critically ill patients undergoing invasive mechanical ventilation. Participants will be randomly assigned to two groups: a control group receiving conventional physical therapy alone and an intervention group receiving conventional physical therapy combined with NMES.

The control group will receive individualized conventional physical therapy, adjusted daily based on each patient's physiological status and following protocols supported by current literature. Interventions may include progressive mobility, such as bed exercises, rolling, sitting at the edge of the bed, standing, chair transfers, and ambulation, as well as respiratory physiotherapy techniques including bronchial hygiene, pulmonary re-expansion, and management of mechanical ventilation. Sessions will last approximately 20 minutes and continue throughout hospitalization, except in cases of clinical contraindications or refusal by the patient/family.

The NMES group will receive the same conventional physical therapy described above, plus NMES applied once or twice daily to both lower limbs for up to 20 consecutive days or until hospital discharge, whichever comes first.

Rectangular electrodes (90 × 50 mm) will be placed bilaterally on the vastus lateralis, vastus medialis, tibialis anterior, hamstrings, and gastrocnemius muscles. If hair interferes with electrode adhesion, the area will be shaved.

NMES will be delivered using the ReCARE® device (Visuri, MG, Brazil) with the following parameters:

Frequency: 60 Hz

Pulse duration: 500 µs

Intensity: adjusted to produce visible muscle contractions during the first two days and, from day three onward, contractions sufficient to generate movement against gravity.

Contraction (on) and relaxation (off) times and the number of contractions will be progressively adjusted according to the 20-day protocol:

Days 1-2: On = 9s, Off = 27s, 16 contractions, 2x/day

Days 3-6: On = 9s, Off = 25s, 26 contractions, 2x/day

Days 6-9: On = 9s, Off = 22s, 60 contractions, 1x/day

Days 10-15: On = 9s, Off = 20s, 70 contractions, 1x/day

Days 16-20: On = 12s, Off = 15s, 70 contractions, 1x/day

NMES sessions will be postponed if the participant exhibits any of the following clinical findings within three hours prior to the session:

Acidosis (arterial pH < 7.25 or venous pH < 7.20)

Hypotension or hypertension (mean arterial pressure < 60 mmHg or > 140 mmHg)

Use of a single vasopressor at >50% of the ICU maximum dose (e.g., dopamine >12.5 µg/kg/min, phenylephrine >2 µg/kg/min, vasopressin ≥0.02 U/min, norepinephrine >1 µg/kg/min)

Use of two vasopressors at ≥40% of the ICU maximum dose

New diagnosis of pulmonary embolism or deep vein thrombosis without anticoagulation for more than 48 hours

Other signs of physiological instability, including temperature <34°C or >41°C, lactate >3.0 mmol/L, creatine kinase >400 U/L, platelet count <20,000/mm³, or suspected muscle inflammation (e.g., rhabdomyolysis, myositis, neuroleptic malignant syndrome, or serotonin syndrome).

This study aims to determine whether NMES, as an early adjunct therapy, can improve recovery and clinical outcomes in critically ill mechanically ventilated patients when combined with conventional physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they are 18 years or older, are under invasive mechanical ventilation (IMV), and are expected to require IMV for more than 48 hours.

Exclusion Criteria:

* Body mass index (BMI) greater than or equal to 35 kg/m²;
* Length of ICU stay longer than 7 ICU-free days or more than 3 continuous days of invasive mechanical ventilation (IMV) before enrollment;
* Known intracranial process (e.g., stroke, intracranial hypertension);
* Neuromuscular disease (e.g., Guillain-Barré syndrome, myasthenia gravis) at ICU admission;
* Inability to speak Portuguese or pre-existing cognitive impairment prior to ICU admission;
* Any condition that prevents neuromuscular electrical stimulation (NMES) treatment or assessment of the primary outcome in both legs (e.g., skin lesions, fractures, or amputation);
* Inability to transfer independently from bed to chair before ICU admission;
* Cardiac arrest as the cause of ICU admission or cardiac arrest before screening;
* Deep vein thrombosis (DVT) or pulmonary embolism (PE) treated for less than 48 hours;
* Pregnant patients;
* Known or suspected malignancy in the legs;
* Any care limitation including a do-not-resuscitate order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Muscle strength assessed by the Medical Research Council (MRC) sum score at ICU discharge | Within 24 hours after ICU discharge
  Muscle strength will be evaluated by trained physiotherapists using the Medical Research Council (MRC) scale, which grades muscle strength from 0 (no contraction) to 5 (normal strength) in key muscle groups, with a maximum total score of 60 points. Muscle weakness is defined as a score below 48 points. This scale provides a standardized method to evaluate muscular recovery during critical illness and hospitalization.

SECONDARY OUTCOMES:
Rectus femoris muscle thickness measured by ultrasound at initiation of invasive mechanical ventilation | within 24 hours after enrollment
  The thickness of the rectus femoris muscle will be measured in millimeters using ultrasound imaging performed by trained professionals, in order to assess muscle morphology.
Rectus femoris pennation angle measured by ultrasound at initiation of invasive mechanical ventilation | within 24 hours after enrollment
  The quadriceps muscle (specifically the rectus femoris) will be evaluated using ultrasound imaging by trained professionals. The pennation angle of the rectus femoris will be measured in degrees to assess muscle architecture.
Rectus femoris pennation angle measured by ultrasound at sedation awakening | Within 24 hours after awakening from sedation in the ICU
  The quadriceps muscle (specifically the rectus femoris) will be evaluated using ultrasound imaging by trained professionals. The pennation angle (in degrees) will be measured. Assessments will be performed when sedation is reduced or stopped to the point that the patient can respond to at least three motor commands (e.g., blink eyes, look at the examiner, stick out tongue, shake head, or raise eyebrows), in order to assess muscle architecture at sedation awakening.
  Unit of Measure: degrees (°)
Rectus femoris muscle thickness measured by ultrasound at sedation awakening | Within 24 hours after awakening from sedation in the ICU
  The quadriceps muscle (specifically the rectus femoris) will be evaluated using ultrasound imaging by trained professionals. Muscle thickness (in millimeters) will be measured. Assessments will be performed when sedation is reduced or stopped to the point that the patient can respond to at least three motor commands (e.g., blink eyes, look at the examiner, stick out tongue, shake head, or raise eyebrows), in order to assess muscle morphology at sedation awakening.
  Unit of Measure: millimeters (mm)
Rectus femoris pennation angle measured by ultrasound at ICU discharge | Within 24 hours after ICU discharge
  The quadriceps muscle (specifically the rectus femoris) will be evaluated using ultrasound imaging by trained professionals. The pennation angle (in degrees) will be measured to assess muscle architecture. Each value will be recorded individually at ICU discharge.
  Unit of Measure: degrees (°)
Rectus femoris muscle thickness measured by ultrasound at ICU discharge | Within 24 hours after ICU discharge
  The quadriceps muscle (specifically the rectus femoris) will be evaluated using ultrasound imaging by trained professionals. Muscle thickness (in millimeters) will be measured to assess muscle morphology. Each value will be recorded individually at ICU discharge.
  Unit of Measure: millimeters (mm)
Rectus femoris pennation angle measured by ultrasound at hospital discharge | From 48 hours to 0 hours before hospital discharge
  The quadriceps muscle (specifically the rectus femoris) will be evaluated using ultrasound imaging by trained professionals. The pennation angle (in degrees) will be measured to assess muscle architecture. Assessments will be performed at hospital discharge.
  Unit of Measure: degrees (°)
Rectus femoris muscle thickness measured by ultrasound at hospital discharge | From 48 hours to 0 hours before hospital discharge
  The quadriceps muscle (specifically the rectus femoris) will be evaluated using ultrasound imaging by trained professionals. Muscle thickness (in millimeters) will be measured to assess muscle morphology. Assessments will be performed at hospital discharge.
  Unit of Measure: millimeters (mm)
Muscle strength assessed by the Medical Research Council (MRC) sum score at awakening from sedation | Within 24 hours after awakening from sedation in the ICU
  Muscle strength will be evaluated by trained physiotherapists using the Medical Research Council (MRC) sum score, which grades muscle strength from 0 (no contraction) to 5 (normal strength) in key muscle groups, with a maximum total score of 60 points. Muscle weakness is defined as a score below 48 points. Assessments will be performed when sedation is reduced or stopped so that the patient can respond to at least three motor commands (e.g., blink eyes, look at examiner, stick out tongue, shake head, raise eyebrows) to assess muscle strength at sedation awakening.
Muscle strength assessed by the Medical Research Council (MRC) sum score at hospital discharge | From 48 hours to 0 hours before hospital discharge
  Muscle strength will be evaluated by trained physiotherapists using the Medical Research Council (MRC) scale, which grades muscle strength from 0 (no contraction) to 5 (normal strength) in key muscle groups, with a maximum total score of 60 points. Muscle weakness is defined as a score below 48 points. Assessments will be performed at three time points: awakening from sedation, ICU discharge, and hospital discharge. This scale provides a standardized method to evaluate muscular recovery during critical illness and hospitalization.
Handgrip strength measured at awakening from sedation in the ICU | Within 24 hours after awakening from sedation in the ICU
  Handgrip strength will be assessed using a handheld hydraulic dynamometer, which measures the maximum force the participant can apply by squeezing the device with their hand. The participant will remain seated with their feet flat on the floor and the arm positioned in a standardized manner to ensure measurement accuracy. Assessments will be performed when sedation is reduced or stopped so that the patient can respond to at least three motor commands (e.g., blink eyes, look at examiner, stick out tongue, shake head, raise eyebrows) to assess muscle.
Handgrip strength measured at ICU discharge | Within 24 hours after ICU discharge
  Handgrip strength will be assessed using a handheld hydraulic dynamometer, which measures the maximum force the participant can apply by squeezing the device with their hand. The participant will remain seated with their feet flat on the floor and the arm positioned in a standardized manner to ensure measurement accuracy.
Handgrip strength measured at hospital discharge | From 48 hours to 0 hours before hospital discharge
  Handgrip strength will be assessed using a handheld hydraulic dynamometer, which measures the maximum force the participant can apply by squeezing the device with their hand. The participant will remain seated with their feet flat on the floor and the arm positioned in a standardized manner to ensure measurement accuracy.
Isometric Knee Extension Strength Assessed at Awakening From Sedation in the ICU | Within 24 hours after awakening from sedation in the ICU
  Isometric knee extension strength will be assessed using a portable dynamometer. Participants will be seated with the knee at a 60-degree angle of flexion and instructed to push the leg forward against the device without moving the joint. This test measures the force generated by the quadriceps while the joint remains still. Assessments will be conducted by trained professionals using standardized procedures. Measurements will be performed when sedation is reduced or stopped so that the patient can respond to at least three motor commands (e.g., blink eyes, look at examiner, stick out tongue, shake head, raise eyebrows) to assess muscle strength at sedation awakening.
Isometric Knee Extension Strength Assessed at ICU Discharge | Within 24 hours after ICU discharge
  Isometric knee extension strength will be assessed using a portable dynamometer. The participant will be seated with the knee positioned at a 60 degree angle of flexion and instructed to push the leg forward against the device without moving the joint. This test measures the force the quadriceps can generate while the joint remains still. The assessment will be conducted by trained professionals using standardized procedures.
Isometric Knee Extension Strength Assessed at Hospital Discharge | From 48 hours to 0 hours before hospital discharge
  Isometric knee extension strength will be assessed using a portable dynamometer. The participant will be seated with the knee positioned at a 60 degree angle of flexion and instructed to push the leg forward against the device without moving the joint. This test measures the force the quadriceps can generate while the joint remains still. The assessment will be conducted by trained professionals using standardized procedures.
Functional capacity assessed by the Six-Minute Walk Test (6MWT) | From 48 hours to 0 hours before hospital discharge
  The six-minute walk test (6MWT) will be conducted by trained physiotherapists to assess functional exercise capacity. The total distance walked in six minutes will be recorded following standardized procedures.
Barthel Index Assessed at Study Enrollment | At baseline (study enrollment)
  Functional independence will be evaluated using the Barthel Index, a questionnaire that measures a patient's ability to perform activities of daily living (ADLs). At study enrollment, the questionnaire will be answered by the patient's family member or primary caregiver to provide a baseline assessment of the patient's functional status prior to ICU admission. The Barthel Index assesses independence in areas such as personal care, mobility, locomotion, and elimination. Each activity is scored based on the patient's level of independence, assistance needed, or dependence. Scores range from 0 to 100 in increments of five, with higher scores indicating greater functional independence.
Barthel Index Assessed at Hospital Discharge | From 48 hours to 0 hours before hospital discharge
  Functional independence will be evaluated using the Barthel Index, a questionnaire that measures a patient's ability to perform activities of daily living (ADLs). The questionnaire assesses independence in areas such as personal care, mobility, locomotion, and elimination. Each activity is scored based on the patient's level of independence, assistance needed, or dependence. Scores range from 0 to 100 in increments of five, with higher scores indicating greater functional independence.
Barthel Index Assessed at 6 Months Post Hospital Discharge | 6 months after hospital discharge
  Functional independence will be evaluated using the Barthel Index, a questionnaire that measures a patient's ability to perform activities of daily living (ADLs). At 6 months post hospital discharge, the patient will be contacted by telephone to complete the questionnaire. The Barthel Index assesses independence in areas such as personal care, mobility, locomotion, and elimination. Each activity is scored based on the patient's level of independence, assistance needed, or dependence. Scores range from 0 to 100 in increments of five, with higher scores indicating greater functional independence.
Duration of invasive mechanical ventilation (IMV) | Within 24 hours after ICU discharge
  The duration of invasive mechanical ventilation (IMV) will be measured from the initiation of IMV until the day of extubation. This duration will be verified and confirmed through review of the patient's medical records.
Ventilator-free days | Within 24 hours after ICU discharge
  The number of days during which the patient was alive and free from invasive mechanical ventilation (IMV) during the ICU stay. This information will be collected from the patient's medical records at hospital discharge.
Length of stay in ICU and hospital | Within 24 hours after hospital discharge
  The total number of days the patient remains admitted in the Intensive Care Unit (ICU) and the hospital during their treatment period. This includes the time from ICU admission until discharge from the hospital. This information will be collected from the patient's medical records at hospital discharge.
Mortality | From hospital admission until death or up to 180 days (6 months) after hospital discharge, whichever occurs first
  The number of deaths occurring among study participants during the hospital stay and within six months after hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Cassiano TEIXEIRA, PhD, Principal Investigator — Hospital Moinhos de Vento
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the study, including the analyzable dataset, will be shared with qualified researchers for academic purposes.
Supporting Information: SAP
Time Frame: Starting 6 months after study completion and available for 5 years
Access Criteria: Qualified researchers affiliated with academic or research institutions will be eligible to access the de-identified individual participant data and supporting documents, including the study protocol and statistical analysis plan. Access will be granted after submission and approval of a research proposal by the study's data sharing committee. Researchers must agree to a data use agreement ensuring confidentiality and appropriate use of the data. Data and documents will be shared via secure data transfer methods.

REFERENCES:
- [Background] Hogrel JY, Benveniste O, Bachasson D. Routine monitoring of isometric knee extension strength in patients with muscle impairments using a new portable device: cross-validation against a standard isokinetic dynamometer. Physiol Meas. 2020 Feb 5;41(1):015003. doi: 10.1088/1361-6579/ab6b49. PMID 31935703
- [Background] Britto RR, Probst VS, de Andrade AF, Samora GA, Hernandes NA, Marinho PE, Karsten M, Pitta F, Parreira VF. Reference equations for the six-minute walk distance based on a Brazilian multicenter study. Braz J Phys Ther. 2013 Nov-Dec;17(6):556-63. doi: 10.1590/S1413-35552012005000122. Epub 2013 Nov 14. PMID 24271092
- [Background] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036
- [Background] Stefanou C, Karatzanos E, Mitsiou G, Psarra K, Angelopoulos E, Dimopoulos S, Gerovasili V, Boviatsis E, Routsi C, Nanas S. Neuromuscular electrical stimulation acutely mobilizes endothelial progenitor cells in critically ill patients with sepsis. Ann Intensive Care. 2016 Dec;6(1):21. doi: 10.1186/s13613-016-0123-y. Epub 2016 Mar 11. PMID 26969168
- [Background] Silva PE, Babault N, Mazullo JB, de Oliveira TP, Lemos BL, Carvalho VO, Durigan JLQ. Safety and feasibility of a neuromuscular electrical stimulation chronaxie-based protocol in critical ill patients: A prospective observational study. J Crit Care. 2017 Feb;37:141-148. doi: 10.1016/j.jcrc.2016.09.012. Epub 2016 Sep 22. PMID 27732921
- [Background] Sachetti A, Carpes MF, Dias AS, Sbruzzi G. Safety of neuromuscular electrical stimulation among critically ill patients: systematic review. Rev Bras Ter Intensiva. 2018 Apr-Jun;30(2):219-225. doi: 10.5935/0103-507X.20180036. PMID 29995088
- [Background] Padte S, Samala Venkata V, Mehta P, Tawfeeq S, Kashyap R, Surani S. 21st century critical care medicine: An overview. World J Crit Care Med. 2024 Mar 9;13(1):90176. doi: 10.5492/wjccm.v13.i1.90176. eCollection 2024 Mar 9. PMID 38633477
- [Background] Paudel R, Trinkle CA, Waters CM, Robinson LE, Cassity E, Sturgill JL, Broaddus R, Morris PE. Mechanical Power: A New Concept in Mechanical Ventilation. Am J Med Sci. 2021 Dec;362(6):537-545. doi: 10.1016/j.amjms.2021.09.004. Epub 2021 Sep 28. PMID 34597688
- [Background] Rodriguez PO, Setten M, Maskin LP, Bonelli I, Vidomlansky SR, Attie S, Frosiani SL, Kozima S, Valentini R. Muscle weakness in septic patients requiring mechanical ventilation: protective effect of transcutaneous neuromuscular electrical stimulation. J Crit Care. 2012 Jun;27(3):319.e1-8. doi: 10.1016/j.jcrc.2011.04.010. Epub 2011 Jun 28. PMID 21715139
- [Background] Nosaka K, Aldayel A, Jubeau M, Chen TC. Muscle damage induced by electrical stimulation. Eur J Appl Physiol. 2011 Oct;111(10):2427-37. doi: 10.1007/s00421-011-2086-x. Epub 2011 Aug 3. PMID 21811767
- [Background] Nakanishi N, Oto J, Tsutsumi R, Yamamoto T, Ueno Y, Nakataki E, Itagaki T, Sakaue H, Nishimura M. Effect of Electrical Muscle Stimulation on Upper and Lower Limb Muscles in Critically Ill Patients: A Two-Center Randomized Controlled Trial. Crit Care Med. 2020 Nov;48(11):e997-e1003. doi: 10.1097/CCM.0000000000004522. PMID 32897665
- [Background] Maffiuletti NA. Physiological and methodological considerations for the use of neuromuscular electrical stimulation. Eur J Appl Physiol. 2010 Sep;110(2):223-34. doi: 10.1007/s00421-010-1502-y. Epub 2010 May 15. PMID 20473619
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Sommers J, Engelbert RH, Dettling-Ihnenfeldt D, Gosselink R, Spronk PE, Nollet F, van der Schaaf M. Physiotherapy in the intensive care unit: an evidence-based, expert driven, practical statement and rehabilitation recommendations. Clin Rehabil. 2015 Nov;29(11):1051-63. doi: 10.1177/0269215514567156. Epub 2015 Feb 13. PMID 25681407
- [Background] Vanhorebeek I, Latronico N, Van den Berghe G. ICU-acquired weakness. Intensive Care Med. 2020 Apr;46(4):637-653. doi: 10.1007/s00134-020-05944-4. Epub 2020 Feb 19. PMID 32076765
- [Background] Hermans G, Van Mechelen H, Clerckx B, Vanhullebusch T, Mesotten D, Wilmer A, Casaer MP, Meersseman P, Debaveye Y, Van Cromphaut S, Wouters PJ, Gosselink R, Van den Berghe G. Acute outcomes and 1-year mortality of intensive care unit-acquired weakness. A cohort study and propensity-matched analysis. Am J Respir Crit Care Med. 2014 Aug 15;190(4):410-20. doi: 10.1164/rccm.201312-2257OC. PMID 24825371
- [Background] Koutsioumpa E, Makris D, Theochari A, Bagka D, Stathakis S, Manoulakas E, Sgantzos M, Zakynthinos E. Effect of Transcutaneous Electrical Neuromuscular Stimulation on Myopathy in Intensive Care Patients. Am J Crit Care. 2018 Nov;27(6):495-503. doi: 10.4037/ajcc2018311. PMID 30385541
- [Background] Kho ME, Truong AD, Zanni JM, Ciesla ND, Brower RG, Palmer JB, Needham DM. Neuromuscular electrical stimulation in mechanically ventilated patients: a randomized, sham-controlled pilot trial with blinded outcome assessment. J Crit Care. 2015 Feb;30(1):32-9. doi: 10.1016/j.jcrc.2014.09.014. Epub 2014 Sep 22. PMID 25307979
- [Background] Fan E, Dowdy DW, Colantuoni E, Mendez-Tellez PA, Sevransky JE, Shanholtz C, Himmelfarb CR, Desai SV, Ciesla N, Herridge MS, Pronovost PJ, Needham DM. Physical complications in acute lung injury survivors: a two-year longitudinal prospective study. Crit Care Med. 2014 Apr;42(4):849-59. doi: 10.1097/CCM.0000000000000040. PMID 24247473
- [Background] Rosa D, Negro A, Marcomini I, Pendoni R, Albabesi B, Pennino G, Terzoni S, Destrebecq A, Villa G. The Effects of Early Mobilization on Acquired Weakness in Intensive Care Units: A Literature Review. Dimens Crit Care Nurs. 2023 May-Jun 01;42(3):146-152. doi: 10.1097/DCC.0000000000000575. PMID 36996359
- [Background] Compston A. Aids to the investigation of peripheral nerve injuries. Medical Research Council: Nerve Injuries Research Committee. His Majesty's Stationery Office: 1942; pp. 48 (iii) and 74 figures and 7 diagrams; with aids to the examination of the peripheral nervous system. By Michael O'Brien for the Guarantors of Brain. Saunders Elsevier: 2010; pp. [8] 64 and 94 Figures. Brain. 2010 Oct;133(10):2838-44. doi: 10.1093/brain/awq270. No abstract available. PMID 20928945
- [Background] Zhu C, Liu B, Yang T, Mei Q, Pan A, Zhao D. [Effect of early rehabilitation physiotherapy on muscle quality and function in critically ill patients]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2018 Jun;30(6):569-572. doi: 10.3760/cma.j.issn.2095-4352.2018.06.013. Chinese. PMID 30009733
- [Background] Xu C, Yang F, Wang Q, Gao W. Effect of neuromuscular electrical stimulation in critically ill adults with mechanical ventilation: a systematic review and network meta-analysis. BMC Pulm Med. 2024 Jan 25;24(1):56. doi: 10.1186/s12890-024-02854-9. PMID 38273243
- [Background] Yurumez B, Metin Y, Atmis V, Karadavut M, Ari S, Gemci E, Yigit S, Ozalp Ates FS, Gozukara MG, Kaplankiran C, Cosarderelioglu C, Yalcin A, Aras S, Varli M. A new possible marker: can pennation angle defined by ultrasound predict the frailty? Aging Clin Exp Res. 2024 Mar 5;36(1):53. doi: 10.1007/s40520-023-02663-w. PMID 38438616
- [Background] De Jonghe B, Bastuji-Garin S, Durand MC, Malissin I, Rodrigues P, Cerf C, Outin H, Sharshar T; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Respiratory weakness is associated with limb weakness and delayed weaning in critical illness. Crit Care Med. 2007 Sep;35(9):2007-15. doi: 10.1097/01.ccm.0000281450.01881.d8. PMID 17855814
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Akar O, Gunay E, Sarinc Ulasli S, Ulasli AM, Kacar E, Sariaydin M, Solak O, Celik S, Unlu M. Efficacy of neuromuscular electrical stimulation in patients with COPD followed in intensive care unit. Clin Respir J. 2017 Nov;11(6):743-750. doi: 10.1111/crj.12411. Epub 2015 Dec 16. PMID 26597394